CLINICAL TRIAL: NCT04701034
Title: Intravenous Immunoglobulin and Prednisolone to Women With Unexplained Recurrent Pregnancy Loss After Assisted Reproductive Technology Treatment: a Randomised, Double-blind, Placebo-controlled Trial
Brief Title: Intravenous Immunoglobulin and Prednisolone for RPL After ART.
Acronym: RPL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Collaborators: Svend Andersen Fonden (Unknown); Beckett Foundation (Other); L.F. Foghts Foundation (Unknown)
Responsible Party: Principal Investigator, Caroline Nørgaard-Pedersen, Dr.med., Aalborg University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CNPOBC2020; 2020-000256-35 (EudraCT Number); U1111-1273-8585 (Other: WHO Universal Trial Number (UTN))
Record Dates: First submitted 2021-01-05; First posted 2021-01-08 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Habitual Abortion; Recurrent Pregnancy Loss; Fertility Disorders; Miscarriage
Keywords: Fertility treatment; In vitro fertilization; Intravenous immunoglobulin; Prednisolone; Recurrent pregnancy loss
MeSH Terms: conditions — Abortion, Habitual; Abortion, Spontaneous | interventions — Immunoglobulins, Intravenous; Prednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: None of the personnel with patient contact will have knowledge to the patient's allocation to active treatment or placebo group. Medicine will be handled at another location and sent to the RPL center masked with universal labels with only name of the patient and study ID number.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active treatment group (Active Comparator): Intravenous immunoglobulin(IVIg) and prednisolone. IVIG is administered at the time of embryo/blastocyst transfer (ET) (5 days before to 2 days after ET) and if the participant becomes pregnant, the infusion (same dose) is repeated in gestational week 5, 6, and 7.
  Participants with pre-pregnancy weight ≤70 kg will receive 25 g immunoglobulin (250 ml), participants with weight 70-85 kg will receive 30 g immunoglobulin (300 ml), and participants with weight ≥85 kg will receive 35 g immunoglobulin (350 ml) at each infusion, which will approximate 0.4 g IVIg per kg body weight.
  Prednisolone, tablets, 5mg. 1 tablet daily started within first 3 days of menstrual cycle and until ET. On the day of ET, the participant will double her dose to 2 tablets daily until a negative pregnancy test, the time of biochemical loss/miscarriage, or pregnancy week 8+0, whichever comes first. Gradual discontinuation four days with one tablet before completing cessation.
  Interventions: Drug: Human Intravenous Immunoglobulins, (Privigen (R), CLS Behring); Drug: Prednisolone Tablets
- Passive treatment group (Placebo Comparator): Human albumin infusion and placebo tablets.
  Human albumin, 5%, (CLS Behring). Participants with pre-pregnancy weight ≤70 kg will receive 250 ml, participants with weight 70-85 kg will receive 300 ml, and participants with weight ≥85 kg will receive 350 ml at each infusion. Administration is planned at the time of ET (5 days before to 2 days after ET) and if the participant becomes pregnant, the infusion is repeated in the same volume in gestational week 5, 6, and 7.
  Placebo tablets: contain 85 mg of lactose monohydrate, 86 mg potato starch, 8.1 mg talc, 3 mg gelatine, and 0.9 mg magnesium stearate. 1 tablet daily started within first 3 days of menstrual cycle and until ET. On the day of ET, the participant will double her dose to 2 tablets daily until a negative pregnancy test, the time of biochemical loss/miscarriage, or pregnancy week 8+0, whichever comes first. Gradual discontinuation four days with one tablet before completing cessation.
  Interventions: Drug: Human Albumin Solution; Drug: Placebo tablet

INTERVENTIONS:
Drug: Human Intravenous Immunoglobulins, (Privigen (R), CLS Behring) — infusion: Initial infusion rate of 0.3 ml/kg BW/hr in about 30 min. If well-tolerated, the infusion rate may gradually be increased to 4.8 ml/kg BW/hr. During the infusion, health care personnel are present to secure immediate action in case of serious AR. Blood pressure and pulse is monitored before, during and after the treatment. In case of anaphylaxis, the treatment is discontinued and the participant is excluded. The hospital ward possess adrenaline 0.1 % solutions ready in case of anaphylaxis.
  Other Names: IVIg
  Arms: Active treatment group
Drug: Prednisolone Tablets — 5 mg before ET and 10 mg after ET until gestational week 8+0
  Arms: Active treatment group
Drug: Human Albumin Solution — Infusion: Initial infusion rate of 0.3 ml/kg BW/hr in about 30 min. If well-tolerated, the infusion rate may gradually be increased to 4.8 ml/kg BW/hr. During the infusion, health care personnel are present to secure immediate action in case of serious AR. Blood pressure and pulse is monitored before, during and after the treatment. In case of anaphylaxis, the treatment is discontinued and the participant is excluded. The hospital ward possess adrenaline 0.1 % solutions ready in case of anaphylaxis.
  Other Names: Albumin infusion
  Arms: Passive treatment group
Drug: Placebo tablet — 1 tablet before ET and 2 tablets after ET until gestational week 8+0
  Arms: Passive treatment group

SUMMARY:
Recurrent pregnancy loss (RPL) affects around 5 % of women in reproductive age. The underlying cause of RPL is most often unknown, probably multifactorial, and no treatment with documented effect on chance of live birth exists. In unexplained cases of RPL, primarily the immune system is hypothesized to play a pivotal, causative role, since autoantibodies and specific human leukocyte antigen (HLA) alleles as well as unbalanced distribution of leucocyte subsets, especially natural killer (NK) cells and T-helper (Th) cells, occurs more frequently in patients with unexplained RPL. For that reason, many treatment regimens used in autoimmune diseases have been tested on RPL patients, as for example prednisolone and intravenous immunoglobulin (IVIg).

IVIg (Privigen) consist of a broad spectrum of structurally and functionally intact IgG antibodies. The mechanism of action is not fully elucidated, but certainly IVIg do help opsonise and neutralize foreign cells and pathogens. Prednisolone support this anti-inflammatory action by suppressing migration of polymorphonuclear leukocytes, and reducing the volume and activity of the immune system and the capillary permeability.

A retrospective, observational pilot study suggested that a combination of prednisone and IVIg in first trimester improves the chance of a live birth in women with RPL after assisted reproductive technologies (ART) (Nyborg et al., 2014).

A randomized controlled study is necessary for determining if this immunomodulatory treatment definitely is effective in patients with unexplained RPL after ART (defined as IVF or ICSI ad FER). Potentially, this study will be able to establish evidence for an effective treatment to women with unexplained RPL after ART, who otherwise have a poor prognosis.

DETAILED DESCRIPTION:
In a randomized, double-blinded, placebo-controlled trial, this study aims to investigate whether treatment with prednisolone and intravenous immunoglobulin (IVIg) before and in early pregnancy improves the chance of a live birth in women undergoing treatment with artificial reproductive technologies (ART) (defined as IVF or ICSI or FER treatment) after previous recurrent pregnancy loss (RPL) after ART.

If an improved live birth rate can be confirmed, the treatment will be the first documented treatment supplement for women with RPL undergoing ART treatment. A treatment with such effect is highly desirable. If the treatment increases the birth rate, it will potentially also improve quality of life and reduce detrimental anxiety and stress symptoms associated with RPL and ART treatment, since the burden (including the number of treatments and the number of losses) will be reduced.

Potential study participants will be identified among patients who are referred to The Center for Recurrent Pregnancy Loss of Western Denmark (in the following called The RPL Center), located at Aalborg University Hospital (AaUH) Denmark.

At the first appointment at The RPL Center, a list of standard health information important for the RPL examination will be collected together with the RPL Center's standard blood sample.

Treatment: The participants will be randomly allocated 1:1 to active immunomodulatory treatment versus placebo treatment (see Arms and Interventions). Study treatment starts on the patient's first day of her menstrual cycle in which her fertility clinic plan to transfer an embryo/blastocyst(s) and continue until a negative pregnancy test, the time of biochemical pregnancy loss/miscarriage or pregnancy week 8+0, whichever comes first.

from first day of cycle and until embryo transfer, one tablet (5mg prednisolone or placebo) per day is taken. First infusion (IVIg or Albumin) is given within 5 workings days before and 2 working days after embryo transfer. On the day of embryo transfer, two tablet per day is taken.

Approximately 14 days after ET, the patient will have a pregnancy test. If positive, the patient will have plasma-hCG measured twice with 1-2 days interval at her local hospital. With adequate increment of plasma-hCG, the patient will be booked for her last 3 infusions in gestational week 5, 6, and 7, and continue tablet intake. If she is not pregnant, study medication will not continue.

On the day of the first infusion treatment and again approximately four weeks later (the day of her third infusion treatment during pregnancy), a study specific blood sample will be taken for our research biobank. In participants who do not achieve pregnancy or have a miscarriage before gestational week 6 (and therefore do not come for the third infusion), we will ask these participants to come for the second blood sample too. The blood samples will be analysed by the Department of Clinical Immunology at AaUH.

In addition, in a separate study performed by the same investigators, a group of 37 healthy females in reproductive age with no prior known pregnancy losses will have one blood sample collected in their luteal phase and analyzed according to the same protocol and will serve as a reference group to the two study groups.

An immediate analysis of the blood sample will quantify NK-cells, B-cells, and T-cell subsets by flow cytometry. Also, a TruCulture analysis for activity of leucocyte subsets will be carried out in 25 patients. The research/future biobank will store frozen serum and plasma for analysis of immune markers including smaller extracellular vesicles.

If the participant is still pregnant after her last infusion of study medicine before week 8+0, she will be offered routine monitoring at The RPL Center at AaUH, at her local fertility clinic, and her local hospital. She will receive a questionnaire 2 weeks after her nuchal scan and 2 weeks after her due date for collection of data regarding her pregnancy, delivery, and perinatal outcome.

Study-relevant data will be collected from medical records, birth records, questionnaires, and the research biobank.

Adverse events will be recorded on all participants from the day of admission and until 6 months after last infusion treatment or until birth of her child if she becomes pregnant. Both adverse events in the participant and her child will be recorded. To support compliance and meticulous reporting of side effects, all participants receive a folder with a list of all known side effects to prednisolone, IVIg and albumin, a diary with boxes to tick of every day the tablet(s) is taken, and a table in which side effects can continuously be noted. According to the child, negative perinatal outcomes (e.g., low birth weight, preterm birth, stillbirth) and malformations will be recorded after birth.

ELIGIBILITY:
Inclusion Criteria:

* Women with ≥ 2 consecutive pregnancy losses (miscarriages or biochemical pregnancies) ≤ completed gestational week 10 after ART with the present partner or with an egg/semen donor*

  * The gestational week of the non-induced pregnancy losses will be based on the date of clinical signs of miscarriage or the fetus' crown-rump-length of a missed abortion measured on the ultrasonic scan detecting the pregnancy loss. If the participant plan to use egg donation in the study cycle, the previous two pregnancy losses must also have happened with the use of egg donation; however, it is not required to use the same egg donor in all three embryo transfers.

Exclusion Criteria:

1. BMI ≥35
2. Age ≥41
3. Significant uterine malformation(s)
4. Known parental balanced chromosomal translocations
5. ≥2 previous pregnancies with fetuses with known abnormal karyotype
6. Patients with IgA deficiency, IgA-autoantibodies or hyperprolinaemia
7. Treatment with medication interacting with prednisolone

   * CYP3A4-inhibitors (fx erythromycin, itraconazole, ritonavir, lopinavir), CYP3A4-inductors (fx phenobarbital, phenytoin og rifampicin), loop diuretics, thiazides, amphotericin B, beta2-agonists, antidiabetics, interleukin-2, somatotropins, anticholinergics and regular treatment with NSAIDs.
8. Patients with moderate/severe hypertension, diabetes mellitus, heart insufficiency, severe mental disorders, Cushing syndrome, myasthenia gravis, ocular herpes simplex, pheochromocytoma, systemic sclerosis, and moderate/severe renal dysfunction.
9. Patients with a clinical or biochemical profile indicating need for heparin or levothyroxine treatment during pregnancy
10. Previous treatment with IVIg
11. Allergy to prednisolone and/or IVIg
12. AMH <4 pmol/L. If transfer of donor egg is planned for her IVF cycle, the AMH value will not be an exclusion criterion.

Ages: 18 Years to 41 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2021-01-28 (Actual); Primary Completion 2024-04-18 (Actual); Study Completion 2024-04-18 (Actual)

PRIMARY OUTCOMES:
A normal live fetus at nuchal scan in ITT population | 12 week after embryo transfer
  The frequency of participants with minimum one apparently normal fetus alive at the time of nuchal scan (approx. week 12) in patients receiving active and placebo treatment, respectively.
  Here, the primary analyses will be undertaken as an intention-to-treat (ITT) analysis, including all participants who were allocated to either active or placebo treatment at the start of the ART cycle, even if they did not receive infusion with IVIg or albumin due to cancellation of embryo/blastocyst transfer.
A normal live fetus at nuchal scan in PP population | 12 week after embryo transfer
  The frequency of participants with minimum one apparently normal fetus alive at the time of nuchal scan (approx. week 12) in patients receiving active and placebo treatment, respectively.
  Here, the primary analyses will be undertaken as a per-protocol (PP) analysis, including patients who were randomized and received the allocated infusion of study medicine at the time of embryo/blastocyst transfer and had this transfer performed.
Live birth rate in ITT population | At delivery
  The frequency of participants with a liveborn (sign of life immediately af delivery >24 weeks) among all randomized participants
Live birth rate in the PP population | At delivery
  The frequency of participants with a liveborn (sign of life immediately af delivery >24 weeks) among all participants who fulfill criteria for PP-analysis
A normal live fetus at nuchal scan among participants who become pregnant after embryo transfer in the ITT population | 12 week after embryo transfer
  The frequency of participants in the ITT population with minimum one apparently normal fetus alive at the time of nuchal scan (approx. week 12) in patients receiving active and placebo treatment, respectively, and who become pregnant after embryo transfer.
A normal live fetus at nuchal scan among participants who become pregnant after embryo transfer in the PP population | 12 week after embryo transfer
  The frequency of participants in the PP population with minimum one apparently normal fetus alive at the time of nuchal scan (approx. week 12) in patients receiving active and placebo treatment, respectively, and who become pregnant after embryo transfer.

SECONDARY OUTCOMES:
Maternal adverse reactions | 9 months after embryo transfer.
  Number of participants with adverse reactions including headache, skin rash, and fever that might be associated to study medicine in the ITT population.
Negative pregnancy test | 9 months after embryo transfer.
  Number of participants with a negative pregnancy test after ET in the ITT population.
Miscarriage rate | Before 24 weeks of gestation
  Number of participants with a miscarriage (defined as any loss before 24 weeks of gestation) among the number of participants becoming pregnant (defined as a rise in serum beta hCG concentration >25 UI/L per transfer) in the ITT population.
Rate of Abnormal karyotype in Miscarried fetuses | Before 24 weeks of gestation
  The frequency of pregnancy losses with unknown or normal karyotype among all participants with a pregnancy loss having an evac. and chromosome typing.
Rate of Stillbirth rate | 9 months after embryo transfer.
  Number of participants with a still birth (defined as fetal death at 24 weeks or more or no sign of life after delivery) among the number of participants becoming pregnant (defined as a rise in serum beta hCG concentration >25 UI/L per transfer) in the ITT population.
Rate of Congenital deformities | 1 week after delivery
  Number of live-born babies with a of congenital deformity among all live-borns in the ITT population.
Rate of Preterm birth | 1 week after delivery
  Number of live-born before 37+0 weeks of gestation among all live-borns in the ITT population.
Rate of Low birth weight (BW) | 1 week after delivery
  Number of live-born with a BW <2500 g among all live-borns in the ITT population.
Rate of Preeclampsia | 1 week after delivery
  Number pregnant participants >24 weeks with hypertension (systolic blood pressure (SBP) greater than or equal to 140 mm Hg or a diastolic blood pressure (DBP) greater than or equal to 90 mm Hg) and proteinuria (>0.3 g per day or urine albumine/creatinine ratio≥ 300 mg/g) among all pregnant participants >24 weeks in the ITT population.
Rate of Gestational diabetes | 1 week after delivery
  Number pregnant participants >24 weeks with gestation diabetes (i.e.efined as an oral glucose challenge test (OGCT) with >9.0 mmol/l 2 hours after oral intake of 75g glucose solution) among all pregnant participants >24 weeks in the ITT population.
Rate of gestational hypertension | 1 week after delivery
  Number pregnant participants >24 weeks with hypertension (i.e. systolic blood pressure (SBP) greater than or equal to 140 mm Hg or a diastolic blood pressure (DBP)) among all pregnant participants >24 weeks in the ITT population.
Rate of abnormal embryonic/fetal karyotype | Before 24 weeks of gestation
  Number of miscarriages with a abnormal embryonic/fetal karyotype among all miscarriages having a karyotype test in the ITT population.
Frequency of a boy | Right after delivery
  The percentage of live births that was a boy

CONTACTS AND LOCATIONS:
Overall Officials: Ole B Christiansen, Principal Investigator — Aalborg University Hospital, Denmark
Locations (1):
- • The Centre for Recurrent Pregnancy Loss of Western Denmark, Department of Obstetrics and Gynaecology, Aalborg University Hospital, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: Yes
The data that will be shared includes (due to the danish regulation) an overview of the data results with means, medians and standard deviations on numbers reported in manuscripts (text, tables, figures, and appendices). If allowed, individual data on these variables will be shared after deidentification together with data dictionary upon request. Sharing will be done after publication and will be available up to 5 years after study end. Study protocol will be available. Data will only be shared with researchers who provide a methodologically sound proposal according to CNP and OBC (the two primary investigators). Proposals should be directed to c.noergaardpedersen@rn.dk. To gain access, data requestors will need to sign a data access agreement.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After results have been published in a manuscript.
Access Criteria: If allowed, individual data on these variables will be shared after deidentification together with data dictionary. Sharing will be done after publication and will be available up to 5 years after study has ended. Study protocol will be available too. Data will only be shared with researchers who provide a methodologically sound proposal according to CNP and OBC (the two primary investigators). Proposals should be directed to c.noergaardpedersen@rn.dk. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Norgaard-Pedersen C, Kesmodel US, Jorgensen MM, Christiansen O. Intravenous immunoglobulin and prednisolone to women with unexplained recurrent pregnancy loss after assisted reproductive technology treatment: a randomised, double-blind, placebo-controlled trial. BMJ Open. 2025 Nov 19;15(11):e106024. doi: 10.1136/bmjopen-2025-106024. PMID 41263919
- [Derived] Norgaard-Pedersen C, Nielsen K, Steffensen R, Eriksen L, Jorgensen MM, Kesmodel US, Christiansen OB. Intravenous immunoglobulin and prednisolone to women with unexplained recurrent pregnancy loss after assisted reproductive technology treatment: a protocol for a randomised, double-blind, placebo-controlled trial. BMJ Open. 2022 Sep 22;12(9):e064780. doi: 10.1136/bmjopen-2022-064780. PMID 36137638